CLINICAL TRIAL: NCT06193512
Title: Efficacy of A Novel RinSe Device to Reduce Oral Bacteria in Intubated IntEnsive CaRe Patients: a Pilot Study (EASIER PILOT)
Brief Title: Efficacy of A Novel RinSe Device to Reduce Oral Bacteria in Intubated IntEnsive CaRe Patients: a Pilot Study
Acronym: EASIER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Swiftsure (Unknown)
Responsible Party: Principal Investigator, Marcelo Gama de Abreu, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23-884
Record Dates: First submitted 2023-11-29; First posted 2024-01-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Oral Bacterial Infection; Mechanical Ventilation Complication

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant, Investigator
Masking Description: Patients and Investigator will be specifically blinded to oral care management whereas the care provider will be unblinded to the oral care management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SwishKit + Oral care treatment as usual (Experimental): SwishKit + Oral care Treatment as usual (TAU)
  Interventions: Device: SwishKit + Oral care treatment as usual
- Oral care treatment as usual (Active Comparator): Oral care Treatment as usual (TAU)
  Interventions: Procedure: Oral care treatment as usual

INTERVENTIONS:
Device: SwishKit + Oral care treatment as usual — SwishKit + Oral care Treatment as usual (TAU) group, instillation of chemical antimicrobial agents care and tooth brushing will be performed as in Oral Care TAU, but SwishKit care will be conducted after other oral care interventions, and prior to instillation of the chemical antimicrobial agent.
  Arms: SwishKit + Oral care treatment as usual
Procedure: Oral care treatment as usual — Oral care will be delivered per standard operating procedure of the ICU, which may include the instillation of chemical agents for the purpose of reducing bacterial load, will be administered at 4-hour intervals, and tooth brushing performed twice daily (morning and evening).
  Arms: Oral care treatment as usual

SUMMARY:
We propose a randomized pilot/feasibility study comparing oral care treatment as usual (TAU) with Swiftsure SwishKit plus oral care TAU on the presence and magnitude of bacterial load in the oropharyngeal space in orotracheally intubated patients. The trial will be conducted with IRB approval and written consent from patient or its legal representative.

DETAILED DESCRIPTION:
Qualifying patients will be assigned on a 1:2 (control : treatment intervention) basis using computer-generated codes and random block sizes without stratification to the following groups:

* Oral care TAU
* Swiftsure SwishKit oral flush plus oral care Treatment as Usual (SK+Oral care TAU)

In the Oral care TAU group, oral care will be delivered per standard operating procedure of the ICU, which may include the instillation of chemical agents for the purpose of reducing bacterial load, will be administered at 4-hour intervals, and tooth brushing performed twice daily (morning and evening). In the SK+Oral care TAU group, instillation of chemical antimicrobial agents care and tooth brushing will be performed as in Oral Care TAU, but SwishKit care will be conducted after other oral care interventions, and prior to instillation of the chemical antimicrobial agent. In both groups, treatment will be conducted for up to 5 days, or until extubation.

Detailed interventions:

Oral care TAU (Treatment as Usual) Standard oral care procedures are designed to help remove microorganisms from mouth surfaces and represent a comprehensive suite of interventions. Oral care provision is codified in a written oral care protocol at the Critical Care unit. The Association of Critical Care Nurses calls for oral care every 2-4 hours. This protocol calls for oral care provision at 4-hour intervals. Oral hygiene will consist of assessment of any plaque buildup on teeth or presence of infection. Brushing and cleaning of the mouth surfaces, followed by administration of a moisturizer to the oral mucosa and lips is required. Oral care includes an assessment of the patient on admission to identify oral health status and self-care deficiencies for further action. Dental plaque removal by brushing the teeth with a soft toothbrush at least twice a day is intended to help remove dental plaque. A toothpaste to assist in breakdown of mucous and biofilm can be administered during brushing. Specific to TAU, nursing will help maintain saliva production to minimize mucositis. The head of the bed will be elevated to at least 30° and positioned to allow secretions to pool in the buccal pocket (especially during tooth brushing and feeding), and the provision of sub-glottic suctioning as needed dependent on mucous production.

SwishKit + Oral care TAU The SwishKit device will be used in accordance with the Operators Manual. The SwishKit device will be inserted into the mouth of the patient by a nurse, and the patient will be properly positioned before use of the device.

A total of 60 mL of 0.9% NaCl will be instilled using three x 20 mL aliquots delivered by syringe (syringe inlet), and immediately evacuated by suction. Upon completion, the SwishKit will be removed and disposed of. The nurse will assure that there is no residual saline or other fluid in the mouth or upper airway, and original position for care resumed.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years or older
* Individual or legally authorized representative consent
* Intubated with an oral endotracheal tube and expected to remain intubated for at least 2 days.

Exclusion Criteria:

* Maxillofacial trauma (current maxillofacial trauma precluding standard oral care techniques)
* Conditions precluding lateral Trendelenburg positioning (e.g., increased intracranial pressure, spinal instability, hemodynamic instability)
* Oropharyngeal injury or infection
* Orofacial edema precluding access for oral care
* Known or anticipated difficult intubation
* Endotracheal cuff air leak that clinicians believe precludes mouth lavage
* Already intubated for more than 24 continuous hours within a week before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bacterial load in the oropharyngeal space | Within 5 days after enrolment.
  Incidence of the presence of bacterial load in the oropharyngeal space from culture and qPCR of the five target pathogens: Enterococcus faecium, Staphylococcus aureus, Klebsiella pneumoniae, Acinetobacter baumannii, Pseudomonas aeruginosa, and Enterobacter spp.

SECONDARY OUTCOMES:
Colony-Forming Units/milliliter (ml) (CFU/ml) | Within 5 days after enrolment.
  Mean colony-forming units/milliliter (ml) (CFU/ml).
16S rRNA sequencing of bacteria | Within 5 days after enrolment.
  16S rRNA sequencing for bacterial identifications and bioinformatics analysis.
Colony-Forming Units/milliliter (ml) (CFU/ml) and 16S rRNA | Within 2 days after enrolment
  Changes in colony-forming units/milliliter (ml) (CFU/ml) and 16S rRNA sequencing between before and after treatment at morning 1 and morning 2.

OTHER OUTCOMES:
Clinician Perception of Treatment Use/Efficacy | Within 5 days after enrolment.
  Qualitatively evaluation of clinician perception of several aspects of the oral care provided by the Swiftsure SwishKit or TAU.
Feasibility aims | Within 5 days after enrolment.
  Qualitatively evaluate 1) procedures related to the timing of the administration of Swiftsure SwishKit oral flush plus oral care TAU; and b) feasibility and methodology of the microbiological sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Gama de Abreu, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No